CLINICAL TRIAL: NCT05581121
Title: PARa-aOrtic LymphAdenectomy in Locally Advanced Cervical Cancer
Acronym: PAROLA
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Claudius Regaud (Other)
Collaborators: ARCAGY/ GINECO GROUP (Other); European Network of Gynaecological Oncological Trial Groups (ENGOT) (Other); Gynecologic Cancer Intergroup (GCIG) (Other); Grupo Español de Investigación en Cáncer de Ovario (Other); Multicenter Italian Trials in Ovarian cancer and gynecologic malignancies (Unknown); Belgian Gynaecological Oncology Group (Other); Swiss GO Trial Group (Network); Institute of Cancer Research, United Kingdom (Other); The Central and Eastern European Gynecologic Oncology Group (Other); Hellenic Cooperative Oncology Group (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 22GENF08
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Cervical Carcinoma; Adenocarcinoma; Adenosquamous Carcinoma
Keywords: Locally advanced cervical cancer; HPV 16+; Stage IIIC1; Radiation therapy; Cisplatin; Para-aortic lymphadenectomy; INTERLACE; KEYNOTE-A18
MeSH Terms: conditions — Uterine Cervical Neoplasms; Adenocarcinoma; Carcinoma, Adenosquamous

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm A (Other): Control arm
  Interventions: Other: Standard treatment: Control arm
- Arm B (Experimental): Experimental arm
  Interventions: Procedure: Experimental arm

INTERVENTIONS:
Other: Standard treatment: Control arm — Standard chemo-radiotherapy and brachytherapy according to EMBRACE II and ESGO/ESTRO recommendations.
  Arms: Arm A
Procedure: Experimental arm — Pre-therapeutic para-aortic lymphadenectomy (by minimally invasive approach) followed by tailored chemo-radiotherapy and brachytherapy. Both traditional laparoscopy or robotically assisted laparoscopy approaches are accepted in the study.
  Arms: Arm B

SUMMARY:
This is an international, multicenter and randomized open-label phase III study designed to demonstrate, in patients with stage IIIC1 cervical cancer, whether para-aortic lymphadenectomy followed by tailored chemoradiation is associated with increased disease-free survival compared to patients staged with FDG-PET/CT only followed by chemoradiation.

The planned sample size is 510; including 200 patients in France.

In this trial, patients will be assigned in one of the two following treatments arms:

* Arm A (control arm): Standard chemo-radiotherapy and brachytherapy according to EMBRACE II and ESGO/ESTRO recommendations.
* Arm B (experimental arm): Pretherapeutic para-aortic lymphadenectomy followed by tailored chemo-radiotherapy and brachytherapy.

Considering the changing standard treatment landscape of locally advanced cervical cancer, both arms (control arm and experimental arm) may also be treated according to the INTERLACE and KEYNOTE-A18 studies, if applicable, at the discretion of the attending physician.

Each patient will be followed up for 5 years.

A cost-utility study will be performed in patients included in France. Other countries could be involved in this specific study. It will assess the incremental cost-utility ratio (cost per QALY gained) of para-aortic lymphadenectomy followed by tailored chemo-radiation in patients with positive PALN compared to patients staged with PET/CT only followed by chemo-radiation.

This study also has ancillary objectives:

* Biologic: To study T cell exhaustion, immune changes during chemoradiation, HPV ctDNA dynamic evolution, and the par-aortic lymph node as a premetastatic niche.
* Radiomics: To study the contribution of radiomics and FDG-PET/CT metabolic parameters to predict para-aortic lymph node involvement and clinical outcome.
* Senti-PAROLA: To evaluate the accuracy (Sensitivity, specificity, positive and negative predictive value) of the para-aortic sentinel lymph node (SPA) for PALN staging, and to evaluate the prognostic value of low volume metastasis of SPA.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years at time of study entry
2. Newly diagnosed histologically proven cervical squamous carcinoma, adenocarcinoma, or adenosquamous tumor
3. FIGO stage IIIC1 (FIGO 2018) cervical cancer with FDG-PET/CT showing FDG-positive pelvic nodes and FDG-negative PALN including equivocal lymph nodes in the common iliac and para-aortic regions. The highest positive lymph node must be located inferior to the common iliac bifurcation in both sides (anatomical level 1).
4. Patients with TNM T stage I-IIIB.
5. FIGO stage IIIC1 cervical cancer by positive pelvic sentinel lymph node from surgical staging (either intraoperative assessment (frozen section) or from final histology - patients are not eligible after radical hysterectomy, and FDG-negative common iliac of para-aortic lymph node on PET/CT (performed before or after SLN procedure)
6. Patient eligible for pelvic radiotherapy and cisplatin-based chemotherapy with a curative intent as confirmed by a multidisciplinary board
7. ECOG performance status < 2 i.e. 0 or 1
8. Life expectancy more than 12 months
9. Pretherapeutic imaging FDG-PET/CT images should be available for central review
10. Prior validation of the surgeon's participation in the study by the Quality Assurance Comity
11. Women should be post-menopaused or willing to accept the use of an effective contraceptive regimen during the treatment period. All non-menopaused women should have a negative pregnancy test within 72 hours prior to study entry.
12. Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment and scheduled visits and examinations including follow up
13. Not applicable since protocol revision V4. Patient participating to other clinical trials including immunotherapy strategies or adjuvant chemotherapy is also eligible for the study. Adjuvant treatment must be decided prior to randomization
14. Signed informed consent
15. Patient affiliated to a Social Health Insurance in France (French patients only).

Exclusion Criteria:

1. Unequivocal positive common iliac or para-aortic lymph nodes at pretherapeutic imaging FDG-PET/CT
2. Negative or equivocal pelvic lymph nodes at pretherapeutic imaging FDG-PET/CT
3. Metastatic disease confirmed by FDG-PET/CT
4. Other histologies than adenocarcinoma, squamous cell carcinoma and adenosquamous carcinoma
5. Contraindication for cisplatin-based chemotherapy
6. Women who received any prior treatment for cervical cancer
7. Prior surgery for the cervical cancer, except for cone procedure and pelvic lymph node staging
8. Previous pelvic radiotherapy
9. History of another primary malignancy except for: Malignancy treated with curative intent and with no known active disease after 5 years, adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease, adequately treated carcinoma in situ (any location) without evidence of disease.
10. Any psychological, familial, geographic or social situation, according to the judgment of investigator, potentially preventing the provision of informed consent or compliance to study procedure
11. Patient who has forfeited his/her freedom by administrative or legal award or who is under legal protection (curatorship and guardianship, protection of justice).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 510 (Estimated)
Dates: Start 2023-12-20 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival (DFS) | 5 years for each patient
  DFS is defined as the time from randomization until first relapse (local, regional, or distant), or death from any cause. Patients still alive at the time of analysis without documented event (including lost to follow-up) will be censored at the last valid disease assessment.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years for each patient
  OS is defined by the delay between randomization and death from any cause. Patients still alive at the time of analysis (including lost of follow-up) will be censored at the last known alive date.
Cancer Specific survival (CSS) | 5 years for each patient
  CSS is defined by the delay between randomization and death from cancer. Patients still alive at the time of analysis (including lost of follow-up) or death from other cause will be censored at the last known alive date and date of death, respectively.
Metastasis Free Survival (MFS) | 5 years for each patient
  MFS is defined as the time from randomization until first distant relapse, or death from any cause. Patients still alive at the time of analysis (including loss of follow-up) without appearance of distant relapse will be censored at the last valid disease assessment.
Para-aortic Free Survival (PAFS) | 5 years for each patient
  PAFS is defined as the time from randomization until para-aortic recurrence, or death from any cause. Patients still alive at the time of analysis (including loss of follow-up) without appearance of para-aortic recurrence will be censored at the last valid disease assessment.
Morbidity and adverse events assessed by the toxicity grading of the National Cancer Institute (NCI-CTCAE v 5.0). | 5 years for each patient
Quality of life will evaluated by the EORTC QLQ-C-30 questionnaire and its cervical cancer module (CXC-24) and the EQ-5D-5L questionnaire. | 5 years for each patient
  The QLQ-C-30 response options are a 4-point Likert scale from "not at all" to "very much" or a seven-point Likert scale from "very poor" to "excellent."The QLQ-CX24 consists of 24 questions including symptom items and sexuality items. The scores/dimensions are: Body image, symptom experience, Sexual/Vaginal Functioning, Lymphedema, Peripheral Neuropathy, Menopausal Symptoms, Sexual Worry, Sexual Activity, sexual enjoyment.The EQ-5D-5L has a descriptive component (composed of 5 dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression) and a visual analogue scale (EQ-VAS). The EQ-5D-5L is translated and validated in French with a utility function calculated on the basis of revealed preferences of French population. The utility-preference approach of the EQ-5D-5L provides a scale with cardinal properties to calculate quality-adjusted life years (QALYs) that are uses in cost-utility analyses.
Cost-utility analysis | 5 years for each patient
  Cost per QALYs gained at 3 year and 5-year follow-up:
  * QALYs gained estimated as the area between the quality-adjusted survival curves of both groups.
  * Utilities are derived from the EQ-5D-5L questionnaire using French weights.
False-negative rate of PET/CT and optional ultrasonography | 3 months post-CRT (Chemo-radiotherapy and brachytherapy) treatment for each patient
  False-negative rate of PET/CT and optional ultrasonography for PALN (Para-Aortic Lymph Node) staging is defined as the ratio of the number of patients PALN+ on para-aortic lymphadenectomy (surgical staging) among the number of patients randomized in the experimental arm (in the overall population and in the subgroup of patients with equivocal lymph nodes).

CONTACTS AND LOCATIONS:
Locations (30):
- France (28):
  - Institut de Cancérologie de l'Ouest, Angers
  - Institut Bergonié, Bordeaux
  - CHU Brest, Brest
  - Centre François Baclesse, Caen
  - Centre Hospitalier Intercommunal de Créteil, Créteil
  - Centre Georges François Leclerc, Dijon
  - Centre Oscar Lambret, Lille
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - Centre Léon Bérard, Lyon
  - Institut Paoli Calmettes, Marseille
  - ICM Val d'Aurelle, Montpellier
  - CHU Nîmes, Nîmes
  - Hôpital Cochin, Paris
  - Hôpital Européen Georges Pompidou, Paris
  - Hôpital Lariboisière Saint Louis, Paris
  - Hôpital Pitié-Salpêtrière, Paris
  - Institut Curie, Paris
  - Hôpital Lyon Sud, Pierre-Bénite
  - Institut Godinot, Reims
  - Centre Henri Becquerel, Rouen
  - Institut Curie Site - Saint Cloud, Saint-Cloud
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Centre Hospitalier Universitaire La Reunion, Saint-Pierre
  - CHRU Strasbourg - ICANS, Strasbourg
  - Institut Universitaire du Cancer Toulouse - Oncopole, Toulouse
  - Chru Tours, Tours
  - Institut Gustave Roussy, Villejuif
- Policlinico Universitario Agostino Gemelli, Roma, Italy
- Hospital Clinic Barcelona, Barcelona, Spain

REFERENCES:
- [Derived] Martinez A, Lecuru F, Bizzarri N, Chargari C, Ducassou A, Fagotti A, Fanfani F, Scambia G, Cibula D, Diaz-Feijoo B, Gil Moreno A, Angeles MA, Muallem MZ, Kohler C, Luyckx M, Kridelka F, Rychlik A, Gerestein KG, Heinzelmann V, Ramirez PT, Frumovitz M, Ferron G, Betrian S, Filleron T, Fotopoulou C, Querleu D; PAROLA Study group. PARa-aOrtic LymphAdenectomy in locally advanced cervical cancer (PAROLA trial): a GINECO, ENGOT, and GCIG study. Int J Gynecol Cancer. 2023 Feb 6;33(2):293-298. doi: 10.1136/ijgc-2022-004223. PMID 36717163